CLINICAL TRIAL: NCT03423095
Title: The Effects of a Motor Imagery Exercise Program on Tongue Strength
Brief Title: Motor Imagery Exercise and Tongue Strength
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Collaborators: James Madison University (Other); Texas Christian University (Other); Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00033331
Record Dates: First submitted 2018-01-15; First posted 2018-02-06 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2018-10

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active Jaw Exercise with Relaxation (Placebo Comparator): Participants randomized to this arm will complete active jaw exercises and visualization relaxation exercise (control group).
  Interventions: Behavioral: Active Jaw Exercise with Relaxation
- Active Tongue Exercise (Active Comparator): Participants randomized to this arm will complete active tongue exercises only.
  Interventions: Behavioral: Active Tongue Exercise
- Active Tongue Exercise + Mental Practice (Experimental): Participants randomized to this arm will complete active tongue exercises and mental practice of tongue exercise via motor imagery.
  Interventions: Behavioral: Active Tongue Exercise + Mental Practice
- Mental Practice Tongue Exercise (Experimental): Participants randomized to this arm will complete mental practice of tongue exercise via motor imagery only.
  Interventions: Behavioral: Mental Practice Tongue Exercise

INTERVENTIONS:
Behavioral: Active Jaw Exercise with Relaxation — This is the control group that will complete exercises unrelated to the primary outcome measures.
  Arms: Active Jaw Exercise with Relaxation
Behavioral: Active Tongue Exercise — This is the active comparator group that will complete exercises already shown to increase tongue strength measures.
  Arms: Active Tongue Exercise
Behavioral: Active Tongue Exercise + Mental Practice — This is an experimental group that will complete active tongue and mental tongue exercises to assess effect on tongue strength measures.
  Arms: Active Tongue Exercise + Mental Practice
Behavioral: Mental Practice Tongue Exercise — This is an experimental group that will complete mental tongue exercises only to assess effect on tongue strength measures.
  Arms: Mental Practice Tongue Exercise

SUMMARY:
This research study is a six-week treatment pilot study to compare the effects of different exercise types on measures of tongue strength and swallowing pressure in typically aging older adults. Typically-aging older adults represent a group "at risk" for dysphagia secondary to sarcopenia of striated musculature important to swallowing. Participants at all study sites will be randomly selected into one of four study exercise groups. At some study sites, the investigators will also determine cortical activation patterns differences during motor execution and motor imagery of tongue exercises between the groups using near-infrared spectroscopy. The results of this study will inform refinement/further development of the mental practice protocol to use with patients with dysphagia in future studies.

DETAILED DESCRIPTION:
Although motor imagery (MI) has not yet been researched in the field of swallowing rehabilitation, the potential benefit is far reaching. Difficulty swallowing, or dysphagia, can occur in people who have a history of stroke, head injury, neurological disease (such as Parkinson's disease, ALS, etc.), and head/neck cancer. A person with dysphagia may have difficulty eating everyday foods and may require an altered diet, such as tube feedings or pureed foods. Because of this, having dysphagia is often associated with increased feelings of isolation and depression. Speech-language pathologists work with people with dysphagia to rehabilitate their swallow, with the goal of reducing their risk of choking and improving their ability to eat normal foods. The use of MI as a way to augment dysphagia rehabilitation has implications for patients who aren't safe to have any food by mouth as well as those who fatigue easily.

This research study is a six-week treatment pilot study to determine the effect of motor imagery for tongue strengthening exercises on measures of tongue strength and swallowing pressure in typically aging older adults. Typically-aging older adults represent a group "at risk" for dysphagia secondary to sarcopenia of striated musculature important to swallowing. Participants at all study sites will be randomly selected into one of four groups: 1) placebo (active jaw open against resistance/close against resistance/lateralize/protrusion exercises with relaxation exercises), 2) active tongue exercises against resistance only, 3) active tongue exercises against resistance + motor imagery of tongue exercises against resistance, and 4) motor imagery of tongue exercises against resistance only. In some participants the investigators will also determine cortical activation patterns differences during motor execution and motor imagery of tongue exercises between the groups using near-infrared spectroscopy. The results of this study will inform refinement/further development of the mental practice protocol to use with patients with dysphagia in future studies.

The research questions are as follows:

1. Does a 6 week treatment of motor imagery tongue exercises with or without active tongue exercise improve tongue strength in healthy older adults compared to a 6 week treatment of placebo exercises and 6 week treatment of active tongue strengthening exercises?
2. Does a 6 week treatment of motor imagery tongue exercises with or without active tongue exercise improve swallowing pressures in healthy older adults compared to a 6 week treatment of placebo exercises and 6 week treatment of active tongue strengthening exercises?
3. Does a 6 week treatment of motor imagery tongue exercises with or without active tongue exercise alter cortical hemodynamic response patterns in healthy older adults compared to a 6 week treatment of placebo exercises and 6 week treatment of active tongue strengthening exercises? (JMU participants only).

The investigators hypothesize, based on previous research, that the group receiving both active and MI treatment will make the most gains in all three measures, followed by the active only group, then the MI only group, then the placebo group (control).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 60-89
* < 3 on EAT-10 (Eating Assessment Tool-10) (part of health questionnaire)
* Mean of ≥2.5 on the KVIQ-10 questions (Kinesthetic and Visual Imagery Questionnaire, short version), a screening questionnaire that assesses a person's motor imagery abilities
* > 24 on MMSE (Mini Mental State Examination), a screening questionnaire that assesses cognitive abilities
* Availability to complete a consecutive 6-week exercise regimen
* Access to reliable transportation to and from study site for in-person experimental sessions
* There are certain conditions that are common to the aging study population we are recruiting which will be acceptable: controlled hypertension and controlled diabetes mellitus

Exclusion Criteria:

* History of diagnosed dysphagia (swallowing disorder)
* History of a seizure(s)
* Current or past problem with pain disorders involving the jaw muscles or joint of the mandible (e.g., TMJ (temporomandibular) disorder or myofacial pain disorder) - these are contraindicated for tongue strengthening exercises
* Presence of oral piercings/oral apparatus that may interfere with tongue exercises
* Medical conditions that would affect oral motor performance (e.g., history of acute or degenerative neurological condition, head/neck cancer), as determined by investigator
* History of a diagnosed dementia or other cognitive impairment
* Uncontrolled high blood pressure

Ages: 60 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-12-19 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Tongue strength change | Change from baseline tongue strength at 6 weeks
  Maximum tongue strength as measured using the Iowa Oral Performance Instrument.

SECONDARY OUTCOMES:
Swallowing pressure change | Change from baseline swallowing pressure strength at 6 weeks
  Regular lingual swallowing pressure as measured using the Iowa Oral Performance Instrument.

OTHER OUTCOMES:
Cortical activation pattern change | Change from baseline tongue relative percent change in oxygenation at 6 weeks
  Patterns relative changes of oxygenation during motor execution and motor imagery of tongue movements will be measured in some participants at the James Madison University study site using near-infrared spectroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Hegyi Szynkiewicz, PhD, Principal Investigator — USF Sarasota-Manatee
Locations (1):
- Sarah Hegyi Szynkiewicz, PhD, CCC-SLP, Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
The privacy and confidentiality of the participants will be maintained. Each participant's identity will be disassociated from the participant's personal data - a subject number will be assigned to each participant upon signing of the informed consent. De-identified data will be shared between universities using a secure and password protected account.
Supporting Information: Study Protocol
Time Frame: De-identified data will be shared from the beginning of enrollment between universities using a password secure Box account and only de-identified data will be kept after the project ends.
Access Criteria: De-identified data will be shared from the beginning of enrollment between universities using a password secure Box account to which all investigators have access.

DOCUMENTS (3):
  • Informed Consent Form (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT03423095/ICF_003.pdf
  • Study Protocol (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/95/NCT03423095/Prot_004.pdf
  • Statistical Analysis Plan (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/95/NCT03423095/SAP_005.pdf